CLINICAL TRIAL: NCT06541392
Title: The Effectiveness of Proper Breakfast Times on Cognitive Function and Health Outcomes Among College Students
Brief Title: The Efficacy of Proper Breakfast Times on Cognitive Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Muhammadiyah Aceh (Other)
Responsible Party: Principal Investigator, Riza Septiani, Medical Doctor, University of Muhammadiyah Aceh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LP4MRiset
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Eating, Time Restricted; Cognitive Change; Blood Pressure; Nutrition, Healthy
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breakfast1 (Experimental): This group will have breakfast time at 6.30 to 7.30 am
  Interventions: Other: breakfast 6.30 am
- Breakfast2 (Experimental): This group will have breakfast time from 7.31 am to 8.31 am
  Interventions: Other: breakfast 7.31 am
- Control (No Intervention): This group will have breakfast time according to their wishes.

INTERVENTIONS:
Other: breakfast 6.30 am — This group will have breakfast time from 6.30 to 7.30 am
  Arms: Breakfast1
Other: breakfast 7.31 am — This group will have breakfast time from 7.31 to 8.31 am
  Arms: Breakfast2

SUMMARY:
The goal of this cluster randomized controlled trial is to learn if a proper breakfast time may increase cognitive function. It will also learn about the effectiveness of proper breakfast time on health outcomes. The main questions it aims to answer are:

Does a proper breakfast time increase cognitive function and health outcomes?

Participants will:

* wake up in the morning at 6 o'clock
* Having breakfast at 6.30 - 7.30 am or 7.31-8.31 am, or having breakfast time according to their wishes.
* Having lunch started at 12.00 pm.

DETAILED DESCRIPTION:
This experimental study uses a Cluster Randomized Controlled Trial non-blinding parallel method design. The objective of this study is to assess the effectiveness of proper breakfast time on cognitive function including the focus on learning and mood among university students. Additionally, the study determines health outcomes such as heart rate, systolic blood pressure, diastolic blood pressure, and macro and micronutrient intake. There are a total of 60 participants from three different faculties. All faculties will be randomly selected and assigned to intervention group 1, intervention group 2, and the control group. Each group consists of 20 participants from each faculty in the university. Intervention Group 1 will have breakfast from 6:30 to 7:30 am, and Intervention Group 2 from 7:31 to 8:31 am. Meanwhile, the control group will continue their preferred breakfast routine. The intervention groups are required to wake up at 6:00 am and have lunch at 12:00 pm.

ELIGIBILITY:
Inclusion Criteria:

* Active student in the year 2024
* Not in medication
* Do not have gastritis or any diseases that require to have breakfast earlier in the morning
* Willing to sign an informed consent
* Have health insurance

Exclusion Criteria:

* Abstain in the education session
* Having emotional and mental health problems
* Students in the final class who are undergoing the thesis writing

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Focus | 8 weeks
  To determine the changes in focus between the groups using the Army alpha test
Mood | 8 weeks
  To determine the changes in mood between the groups using the profile of moods state (POMS) questionnaire

SECONDARY OUTCOMES:
Systolic blood pressure | 8 weeks
  To determine the changes in systolic blood pressure between the groups using the sphygmomanometer
Diastolic blood pressure | 8 weeks
  To determine the changes in diastolic blood pressure between the groups using the sphygmomanometer
Heart rate | 8 weeks
  To determine the changes in heart rate between the groups using the sphygmomanometer
macro nutrition intake | 8 weeks
  To determine the changes in macro nutrition intake between the groups using the 3-day food record
micro-nutrition | 8 weeks
  To determine the changes in micro-nutrition intake between the groups using the 3-day food record

CONTACTS AND LOCATIONS:
Overall Officials: Riza Septiani, Ph.D, Principal Investigator — University of Muhammadiyah Aceh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno-Aznar LA, Vidal Carou MDC, Lopez Sobaler AM, Varela-Moreiras G, Moreno Villares JM. [Role of breakfast and its quality in the health of children and adolescents in Spain]. Nutr Hosp. 2021 Apr 19;38(2):396-409. doi: 10.20960/nh.03398. Spanish. PMID 33724048
- [Background] Baharuddin D, Said MA, Majid HA. Protocol For Intervention Study In Reducing Elevated Blood Pressure Through Intermittent Fasting. J Pak Med Assoc. 2023 Nov;73(11):2171-2176. doi: 10.47391/JPMA.7748. PMID 38013523
- [Result] Crabtree DR, Holliday A, Buosi W, Fyfe CL, Horgan GW, Johnstone AM, On Behalf Of The Full Health-Study Group. The Acute Effects of Breakfast Drinks with Varying Protein and Energy Contents on Appetite and Free-Living Energy Intake in UK Older Adults. Geriatrics (Basel). 2022 Jan 30;7(1):16. doi: 10.3390/geriatrics7010016. PMID 35200521
- [Result] Dalgaard LB, Kruse DZ, Norup K, Andersen BV, Hansen M. A dairy-based, protein-rich breakfast enhances satiety and cognitive concentration before lunch in overweight to obese young females: A randomized controlled crossover study. J Dairy Sci. 2024 May;107(5):2653-2667. doi: 10.3168/jds.2023-24152. Epub 2023 Dec 21. PMID 38135050
- [Result] Xian X, Wang C, Yu R, Ye M. Breakfast Frequency and Sleep Quality in College Students: The Multiple Mediating Effects of Sleep Chronotypes and Depressive Symptoms. Nutrients. 2023 Jun 8;15(12):2678. doi: 10.3390/nu15122678. PMID 37375582